CLINICAL TRIAL: NCT00780351
Title: Pharmacokinetics and Dosing of Vancomycin in Sustained Low Efficiency Daily Hemodiafiltration (SLEDD-f)
Brief Title: Dosing Vancomycin in Patients on Sustained Low Efficiency Daily Hemodiafiltration (SLEDD-f)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Fe-Lin L Wu, Director, Department of Pharmacy, National Taiwan University Hospital
Other Study IDs: 200705036M
Record Dates: First submitted 2008-03-05; First posted 2008-10-27 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Acute Renal Failure
Keywords: vancomycin, SLEDD-f
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SLEDD-f, vanco: Surgical ICU patients who is on slow low efficiency daily hemodiafiltration (SLEDD-f) and requires vancomycin therapy
  Interventions: Device: sustained low efficiency daily hemodiafiltration (SLEDD-f)

INTERVENTIONS:
Device: sustained low efficiency daily hemodiafiltration (SLEDD-f) — vancomycin 15mg/kg IV infusion on day 1 from 6PM to 8PM. Start SLEDD-f on day 2 from 9AM to 5PM.

SUMMARY:
1. Sustained low efficiency daily hemodiafiltration(SLEDD-f) is a kind of renal replacement therapy with high-flux dialyser membrane (helixone).
2. The pore size of helixone is larger than most antibiotics, and vancomycin is supposed to be removed during dialysis.
3. Our study wants to find the amount of vancomycin removed during SLEDD-f, and try to find the most appropriate dose regimen for this kind of patients.

DETAILED DESCRIPTION:
Vancomycin is the most important antibiotic in the treatment of resistant G(+) bacteria infections. Close monitor of serum level is important to ensure its safety and effectiveness. So far there is not enough data to support the optimal dose regimen of vancomycin in patients on SLEDD-f. In this study, we draw blood levels between 2 doses of vancomycin to determine the pharmacokinetic parameters of vancomycin and fraction removed by SLEDD-f so as to determine the most appropriate dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Acute renal failure of any cause
* Use SLEDD-f as renal replacement therapy
* Priscribe vancomycin for a known or suspected infection

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-10; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The amount of vancomycin removed during one course of SLEDD-f | 8 hr (during one course of SLEDD-f)
The pharmacokinetics and dosing regimen of vancomycin in patients on SLEDD-f. | 26 hr

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin L Wu, MSCP, Ph.D., Principal Investigator — School of pharmacy, Graduate institute of clinical pharmacy, Department of Pharmacy of National Taiwan University Hospital, College of Medicine, National Taiwan University; Wen-Je Ko, MD, PhD, Principal Investigator — Department of Surgery, National Taiwan University Hospital, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan